CLINICAL TRIAL: NCT06834568
Title: Tandem Freedom - Feasibility Trial 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0020402
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; T1D; Tandem; t:slim X2; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Tandem Freedom (Experimental): After a one week run-in period with Control-IQ technology, participants will use the Tandem Freedom system for one partial day with user initiated mealtime insulin boluses and three days without user initiated mealtime insulin boluses in a supervised hotel setting.
  Participants will also perform exercise challenges.
  Interventions: Device: t:slim X2 insulin pump with Tandem Freedom Algorithm

INTERVENTIONS:
Device: t:slim X2 insulin pump with Tandem Freedom Algorithm — t:slim X2 insulin pump with Tandem Freedom System consists of the Tandem t:slim X2 insulin pump and the Freedom algorithm embedded in the pump. Participants will also use the Dexcom G6 continuous glucose monitoring system.

SUMMARY:
This feasibility study is a prospective, single arm study evaluating the Tandem Freedom system in adults with type 1 diabetes. Existing Control-IQ technology users will use Control-IQ technology at home for a one week run-in, then will use Tandem Freedom in a supervised hotel setting.

DETAILED DESCRIPTION:
After a one week Control-IQ run-in at home, 10 adults who are existing Control-IQ users with type 1 diabetes will use the Tandem Freedom System for 4 nights: 1 day with boluses, and 3 days without boluses, in a supervised hotel setting. Participants will perform exercise challenges. The primary outcome is safety events. CGM time in ranges will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Diagnosis of type 1 diabetes for at least 1 year
* Current Control-IQ user, having been prescribed Control-IQ for at least 3 months
* HbA1c ≤10%, recorded in the last 3 months
* Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol, including performing the weekend hotel observed setting portion of the study.
* Willing to use only aspart (novorapid) or lispro (humalog) insulin with the study pump, with no use of long-acting basal insulin injections, or inhaled insulin with the study pump.

Exclusion Criteria:

* More than 1 episode of diabetic ketoacidosis (DKA) in the past 6 months
* More than 1 episode of severe hypoglycemia (needing assistance) in the past 6 months
* Inpatient psychiatric treatment in the past 6 months
* For Female: Currently pregnant or planning to become pregnant during the time period of study participation

  1. A negative pregnancy test will be required for all females of child-bearing potential
  2. Counseling on appropriate birth control options will be provided to all females of child-bearing potential
* Concurrent use of any non-insulin glucose-lowering agent, other than metformin (for example, GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
* Hemophilia or any other bleeding disorder
* Hemoglobinopathy
* History of heart, liver, lung or kidney disease determined by investigator to interfere with the study
* History of allergic reaction to Humalog or Novorapid
* Use of any medications determined by investigator to interfere with study
* Significant chronic kidney disease (which could impact CGM accuracy in investigator's judgment) or hemodialysis
* Concurrent use of any medication that could interfere with the study CGM, such as hydroxyurea
* History of adrenal insufficiency
* History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not appropriately treated
* History of gastroparesis
* A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
* Participation in another pharmaceutical or device trial at the time of enrollment or anticipated for during the time period of study participation
* Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Study Director — Tandem Diabetes Care, Inc.
Locations (1):
- University of Otago, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilkinson TM, de Bock MI, Meier R, Hurd S, Sasson-Katchalski R, Trahan A, Rueda JR, Sherer N, Stephens M, Meyer B, Gantulga D, Rackow S, D'Souza EW, Briggs P, Corbett JP, Ulrich TR, Pinsker JE. Fully Closed-Loop Insulin Delivery with High-Carbohydrate and High-Fat Meals Using the Tandem Freedom System. J Diabetes Sci Technol. 2025 Nov 14:19322968251389966. doi: 10.1177/19322968251389966. Online ahead of print. PMID 41236930

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tandem Freedom
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (19.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  New Zealand European | 8
  Maori | 1
  Dutch | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Severe Hypoglycemia Events
Description: Number of Participants with One or More Severe Hypoglycemia Events (with cognitive impairment such that assistance of another individual is needed for treatment)
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
Participants
  Control-IQ Run-in Period (7 days) | 0
  Tandem Freedom (3 days) | 0

2. Primary Outcome: Number of Participants With One or More Diabetic Ketoacidosis Events
Description: Number of Participants with One or More Diabetic Ketoacidosis events
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
Participants
  Control-IQ Run-in Period (7 days) | 0
  Tandem Freedom (3 days) | 0

3. Secondary Outcome: Percent Time <54 mg/dL
Description: CGM measured percent time <54 mg/dL
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-in Period (7 days) | 0.4 [0.2 to 1.1]
  Tandem Freedom (3 days) | 0.0 [0.0 to 0.0]

4. Secondary Outcome: Percent Time <70 mg/dL
Description: CGM measured percent time <70 mg/dL
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-in Period (7 days) | 1.8 [0.8 to 3.0]
  Tandem Freedom (3 days) | 0.4 [0.0 to 0.8]

5. Secondary Outcome: Percent Time in Range 70 - 180 mg/dL
Description: CGM measured percent time in range 70 - 180 mg/dL
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-in Period (7 days) | 56.3 [50.9 to 64.0]
  Tandem Freedom (3 days) | 61.0 [58.9 to 73.0]

6. Secondary Outcome: Percent Time in Range > 180 mg/dL
Description: CGM measured percent time in range > 180 mg/dL
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-in Period (7 days) | 41.8 [34.0 to 47.5]
  Tandem Freedom (3 days) | 38.2 [27.0 to 40.6]

7. Secondary Outcome: Percent Time in Range > 250 mg/dL
Description: CGM measured percent time in range > 250 mg/dL
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-in Period (7 days) | 15.0 [12.1 to 18.6]
  Tandem Freedom (3 days) | 5.6 [4.9 to 12.6]

8. Secondary Outcome: Percent Time in Range 70 - 140 mg/dL
Description: CGM measured percent time in range 70 - 140 mg/dL
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
percentage of time
  Control-IQ Run-in Period (7 days) | 33.8 [30.0 to 46.1]
  Tandem Freedom (3 days) | 42.5 [37.9 to 48.6]

9. Secondary Outcome: Mean Glucose (mg/dL)
Description: CGM measured mean glucose (mg/dL)
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: Median of mean glucose values (mg/dL)
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
Median of mean glucose values (mg/dL)
  Control-IQ Run-in Period (7 days) | 178.3 [164.6 to 184.7]
  Tandem Freedom (3 days) | 166.9 [153.3 to 168.0]

10. Secondary Outcome: Glucose Coefficient of Variation (%)
Description: CGM measured Coefficient of Variation (%)
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: Percentage of variation
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
Percentage of variation
  Control-IQ Run-in Period (7 days) | 0.4 [0.3 to 0.4]
  Tandem Freedom (3 days) | 0.3 [0.3 to 0.4]

11. Secondary Outcome: Glucose Standard Deviation (mg/dL)
Description: CGM measured Standard Deviation (mg/dL)
Time Frame: Control-IQ Run-in Period (7 days), Tandem Freedom (3 days)
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Tandem Freedom
Number analyzed (Participants) | 10
mg/dL
  Control-IQ Run-in Period (7 days) | 67.8 [61.0 to 70.2]
  Tandem Freedom (3 days) | 51.3 [45.5 to 64.2]

ADVERSE EVENTS:
Time Frame: 10 days
Groups:
- Run-in Period: One week run-in period with Control-IQ technology.
- Tandem Freedom: Participants will use the Tandem Freedom system for one partial day with user initiated mealtime insulin boluses and three days without user initiated mealtime insulin boluses in a supervised hotel setting. Participants also performed exercise challenges.
Arm/Group | Run-in Period | Tandem Freedom
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period (N=10) | Tandem Freedom (N=10)
Superficial burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Left forearm superficial burn while cooking
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT06834568/Prot_SAP_000.pdf